CLINICAL TRIAL: NCT03556072
Title: If Different Types of Periampullary Diverticula Affect ERCP Cannulation?
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Xun Li, professor，head of surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: PAD affects ERCP cannulation
Record Dates: First submitted 2018-06-02; First posted 2018-06-14 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Intubation;Difficult
Keywords: ERCP; periampullary diverticula; difficulty cannulation; complication; biliary disorder
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intradiverticular papilla (IDP) group: Routine ERCP, recording the endoscopic procedures and observing the intra- and post-operative parameters
  Interventions: Other: Routine ERCP
- Juxtapapillary diverticulum (JPD) group: Routine ERCP, recording the endoscopic procedures and observing the intra- and post-operative parameters
  Interventions: Other: Routine ERCP

INTERVENTIONS:
Other: Routine ERCP

SUMMARY:
To study the influence of different types of periampullary diverticulum(PAD) on ERCP difficult cannulation and postoperative complications.

DETAILED DESCRIPTION:
Periampullary diverticula (PAD) are extraluminal out-pouching of the duodenum mucosa often occurring within a radius of 2-3 cm from the ampulla of Vater or hepatopancreatic ampulla. More PAD cases have been identified over recent years, and it's generally believed that up to 27% of elderly cases may have PAD. Several classifications of PAD have been proposed, and the most commonly used distinguishes intraluminal and extraluminal diverticula. Recent studies suggest that PAD is a risk factor for the development of bile duct diseases, and it may cause endoscopic retrograde cholangiopancreatography (ERCP) procedures to fail, but some other studies have come to the opposite conclusion.

During ERCP procedures, the investigators found that different types of PAD seem to have some differences in the size of the diverticulum, difficulty in intubation, and complications. The investigators plan to this retrospectively study collecting 4 years of cases to evaluate the clinical features of different types of PAD in terms of difficult cannulation and complications.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old ERCP patients
* With native papilla

Exclusion Criteria:

* Unwillingness or inability to consent for the study
* Coagulation dysfunction (INR> 1.5) and low peripheral blood platelet count (<50×10^9 / L) or using anti-coagulation drugs
* Previous ERCP
* Prior surgery of Bismuth Ⅱ, Roux-en-Y and Cholangiojejunostomy
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage or perforation, severe liver disease(such as decompensated liver cirrhosis, liver failure and so on), septic shock
* Biliary-duodenal fistula confirmed during ERCP
* Pregnant women or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-90 years old patients with ERCP indications
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Difficulty cannulation | 1 month
  The inability to achieve selective biliary cannulation by the standard ERCP technique within 10 minutes or 5 attempts or failure of access to the major papilla.

SECONDARY OUTCOMES:
Diameter of diverticulum | 1 month
  Maximum diameter of PAD observed during ERCP
Diameter of common bile duct | 1 month
  Maximum diameter of common bile duct observed during ERCP
X-ray exposure time | 1 month
  The total radiography time during ERCP
Pancreatic duct insertion times | 1 month
  Times of any accessories goes into the pancreatic duct, no matter how depth
Post-ERCP pancreatitis | 1 month
  Upper abdominal pain with serum amylase elevation more than 3 times after the procedure
Perforation | 1 month
  CT scan shows retroperitoneal space fluid or gas
Acute cholangitis | 1 month
  Intermittent chills and fever after ERCP
Operation time | 1 month
  From successful biliary intubation to end of operation
Secondary treatment rate | 1 month
  Some patients require secondary treatment, including management of primary diseases and complications
Hospital stay | 1 month
  Length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Xun Li, M.D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lobo DN, Balfour TW, Iftikhar SY. Periampullary diverticula: consequences of failed ERCP. Ann R Coll Surg Engl. 1998 Sep;80(5):326-31. PMID 9849331
- [Result] Cappell MS, Mogrovejo E, Manickam P, Batke M. Endoclips to facilitate cannulation and sphincterotomy during ERCP in a patient with an ampulla within a large duodenal diverticulum: case report and literature review. Dig Dis Sci. 2015 Jan;60(1):168-73. doi: 10.1007/s10620-014-3321-1. Epub 2014 Aug 20. No abstract available. PMID 25138902
- [Result] Kim KY, Han J, Kim HG, Kim BS, Jung JT, Kwon JG, Kim EY, Lee CH. Late Complications and Stone Recurrence Rates after Bile Duct Stone Removal by Endoscopic Sphincterotomy and Large Balloon Dilation are Similar to Those after Endoscopic Sphincterotomy Alone. Clin Endosc. 2013 Nov;46(6):637-42. doi: 10.5946/ce.2013.46.6.637. Epub 2013 Nov 19. PMID 24340257
- [Result] Katsinelos P, Chatzimavroudis G, Tziomalos K, Zavos C, Beltsis A, Lazaraki G, Terzoudis S, Kountouras J. Impact of periampullary diverticula on the outcome and fluoroscopy time in endoscopic retrograde cholangiopancreatography. Hepatobiliary Pancreat Dis Int. 2013 Aug;12(4):408-14. doi: 10.1016/s1499-3872(13)60063-6. PMID 23924499
- [Result] Tyagi P, Sharma P, Sharma BC, Puri AS. Periampullary diverticula and technical success of endoscopic retrograde cholangiopancreatography. Surg Endosc. 2009 Jun;23(6):1342-5. doi: 10.1007/s00464-008-0167-7. Epub 2008 Sep 26. PMID 18818967